CLINICAL TRIAL: NCT07105020
Title: iCCARE Project #4: Grounded Theory Study of the Social Determinants of Migrant Health Factors Impacting Prostate Cancer Care and Survivorship Among Sub-Saharan African and Caribbean Immigrant Men Diagnosed With Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0229
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theory Study of the Black Immigrant using a SDOH Model (Experimental): Participants will be recruited by utilizing the MD Anderson Cancer Registry
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — Interviews will be conducted in person, over the phone, or via Zoom.

SUMMARY:
This trial is aimed to better understand the impact of migration history on the quality of life of Black immigrant CaP survivors (both SSAI and CI). We will illuminate the full range of racial, social, environmental, behavioral, and structural factors associated with the Black immigrant experience in the US using a SDOH model.

DETAILED DESCRIPTION:
Primary Objective:

ELIGIBILITY:
Inclusion Criteria:

* be male adults (≥18 years old)
* Self-identify as CI and SSAI
* Self-identify as Black or African American
* Have been diagnosed with CaP within the last 10 years
* Have a U.S. address
* Can read and write in English

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org